CLINICAL TRIAL: NCT03984877
Title: Impact of Cardiac Amyloidosis on Patients With Severe Aortic Stenosis Who Undergo Transcatheter Aortic
Brief Title: Impact of Amyloidosis on TAVI Patients
Acronym: AMY-TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Javier López Pais (Other)
Responsible Party: Sponsor-Investigator, Javier López Pais, Sponsor-Investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Other Study IDs: AMY-TAVI
Record Dates: First submitted 2019-01-22; First posted 2019-06-13 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Valve Stenoses, Aortic; Amyloidosis Cardiac
Keywords: TAVI; Aortic Stenosis; Cardiac amyloidosis
MeSH Terms: conditions — Aortic Valve Stenosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amyloidosis: TAVI patients with diagnosis of amyloidosis
  Interventions: Diagnostic Test: Diagnosis of amyloidosis
- Non-Amyloidosis: TAVI patients without diagnosis of amyloidosis
  Interventions: Diagnostic Test: Diagnosis of amyloidosis

INTERVENTIONS:
Diagnostic Test: Diagnosis of amyloidosis — Scintigraphy and protein electrophoresis

SUMMARY:
To analyze the prevalence and impact on the prognosis of amyloidosis due to transthyretin in patients with severe aortic stenosis who undergo percutaneous aortic valve implantation.

DETAILED DESCRIPTION:
Type and design of the study: Multicentric, prospective cohort, observational.

Number and characteristics of the patients: 321 patients to whom TAVI has been implanted due to severe degenerative AS.

Duration of the study

* Recruitment period: All consecutive patients undergoing a non-invasive diagnostic study of amyloidosis (scintigraphy with technetium pyrophosphate99 and blood protein electrophoresis) will be recruited before discharge, in centers with proven experience, will accept non-invasive diagnosis with resonance) and have an implanted percutaneous aortic prosthesis for severe aortic stenosis.
* Follow-up period: clinical and echocardiographic follow-up will be carried out before discharge, in consultation at three, six, twelve and twenty-four months.

Inclusion: 1 year

Follow up: 2 years

Data analysis: 6 months

Total: 3 years and 6 months

Events

* Main event: cardiovascular events (cardiovascular death, stroke, infarction)
* Secondary events: death from any cause, readmission due to heart failure, pacemaker implantation, functional class evaluation

Countries and participating centers: Various Spanish and international centers will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve replacement with a percutaneous prosthesis due to severe aortic stenosis after evaluation by the Heart Team.
* Ability to understand and sign informed consent.
* They do not meet any of the exclusion criteria.

Exclusion Criteria:

* Death as a complication of the procedure during hospitalization.
* Associated mitral valve disease requiring intervention
* TAVI valve-in-valve implant.
* Does not sign informed consent.

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients of legal age, recruited in the hospitalization area or from outpatient clinics, who meet the following requirements: diagnosis of severe aortic stenosis by conventional echocardiographic criteria (maximum speed> 4m / s, medium transvalvular gradient> 40mmHg, area <1cm2).
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
  Survival after TAVI of patients with amyloidosis

SECONDARY OUTCOMES:
Pacemaker requirements | 15 days
  Number of patients with amyloidosis who received pacemaker after TAVI.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ramón Gonzalez Juantey, M.D. Ph.D., Study Chair — Complexo Hospitalario Universitario de Santiago de Compostela
Locations (1):
- Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03984877/Prot_SAP_000.pdf